CLINICAL TRIAL: NCT01616017
Title: Comparison of Cardiac Output Measured by Ultrasound Dilution Method and Pulmonary Artery Thermodilution Technique
Status: Completed | Type: Observational
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-G-COstatus-11A-H; R44HL061994 (NIH)
Record Dates: First submitted 2012-05-29; First posted 2012-06-11 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Cardiac Disease; Post Surgery Patients
Keywords: Cardiac output; ultrasound dilution; thermodilution
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Cardiac output (CO) is an important hemodynamic variable in the management of critically ill patients. The pulmonary artery catheter (PAC) requires invasive techniques with potential complications and there is increasing interest in less invasive methods of measuring CO. This study is designed to compare CO values from PAC thermodilution (COTD) and ultrasound dilution (COUD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Presence of arterial catheter plus central venous pressure monitor and pulmonary artery catheter for hemodynamic monitoring.

Exclusion Criteria:

* Age < 18 years of age
* Patients with structurally abnormal heart (e.g. shunt) (confirmed by history taking)
* Patients who have heparin allergy. (Confirmed by history taking)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age ≥ 18 years of age Presence of arterial catheter plus central venous pressure monitor and pulmonary artery catheter for hemodynamic monitoring.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Compare Cardiac Output Measurements | During the stay in the ICU with in situ catheters (expected avg 3 days)
  To compare CO measured by ultrasound dilution method (COUD) and pulmonary artery thermodilution technique (COTD) in SICU (Surgical Intensive Care Unit) patients.

CONTACTS AND LOCATIONS:
Locations (1):
- The Queen's Medical Center, Honolulu, Hawaii, United States